CLINICAL TRIAL: NCT01875042
Title: Does Transcutaneous Electrical Nerve Stimulation (TENS) Affect Pain and Function in Patients With Osteoarthritis of the Knee? ETRELKA, a Randomised Controlled Trial
Brief Title: Effect of Transcutaneous Electrostimulation (TENS) on Pain and Physical Function in Patients With Knee Osteoarthritis
Acronym: ETRELKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Arco Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 118/11
Record Dates: First submitted 2013-05-30; First posted 2013-06-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TENS (Experimental): Transcutaneous Electrical Nerve Stimulation
  Interventions: Device: TENS
- Sham TENS (Sham Comparator): Sham Transcutaneous Electrical Nerve Stimulation
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation
  Arms: TENS
Device: Sham TENS — Sham Transcutaneous electrical nerve stimulation
  Arms: Sham TENS

SUMMARY:
The proposed study is a multi-center, randomized, double blind (patient and assessor), sham controlled clinical trial using a parallel 2 group design recruiting 220 patients of at least 18 years of age. The investigators will include patients presenting with clinically and radiologically diagnosed knee OA according to the criteria of the American College of Rheumatology, who experienced knee pain lasting for at least six months, and were diagnosed with radiographic severity of ≥ 2 on the Kellgren-Lawrence grading system or had one or more of the following signs and symptoms in the knee; restricted range of motion, pain in motion, crepitations, morning stiffness. Patients will be randomly allocated to receive TENS or sham TENS for 3 weeks.

DETAILED DESCRIPTION:
Background

Osteoarthritis (OA) is the most common arthritic condition, which is one of the leading causes of disability in adults. Currently, no treatment can stop or reverse the progressive joint degeneration caused by OA. Most clinical interventions aim to improve pain and physical function. Transcutaneous electrical nerve stimulation (TENS) is widely used in the management of knee OA to relieve osteoarthritic pain and facilitate the performance of therapeutic activities in order to maintain or improve physical function. Although its use is widespread, the available evidence is of questionable quality. An adequately sized and well conducted randomized controlled trial (RCT) investigating the effectiveness and safety of TENS as treatment modality for knee OA is warranted to assist clinicians and policy makers to make decisions that are based on high-quality evidence, ultimately optimizing delivery of health-care in knee OA.

Objective

To determine TENS safety and effectiveness on pain and physical function compared to sham TENS in patients with knee OA.

Methods

Multi-center, randomized, double blind (patient and assessor), sham controlled clinical trial using a parallel 2 group design. Patients will be randomly allocated to receive TENS or sham TENS for 3 weeks. Informed consent of eligible patients will be obtained prior to randomization. Patients will be assigned on a 1:1 basis to the TENS or sham TENS group. Randomization will be centralized using randomization software and an electronic randomization form, generated by the trial coordinating centre (CTU Bern). Patients will be randomized once demographic data and selection criteria are completed by the recruiting physician in an electronic form. Randomization will be stratified according to treatment centre, TENS naivety and clinical severity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of at least 18 years of age
* Clinical or radiological diagnosis of knee OA according to the criteria of the American College of Rheumatology
* Knee pain lasting for six months or longer
* Radiographic evidence of at least one osteophyte at the tibiofemoral joint (Kellgren-Lawrence grade ≥ 2) or one or more of the following signs and symptoms in the knee; restricted range of motion, pain in motion, crepitations, morning stiffness
* Written informed consent

Exclusion Criteria

* Patients diagnosed with rheumatoid arthritis or other musculoskeletal diseases affecting lower extremities
* Relevant effusion in the index knee
* Known current or remittent cancer
* Carry cardiac pacemaker or defibrillator in situ
* Knee surgery in previous 6 months
* Received treatment with arthrocentesis
* Intra-articular injection of steroids in previous 3 months
* Inability to understand instructions or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
WOMAC pain subscale | End of treatment (at 3 weeks)

SECONDARY OUTCOMES:
WOMAC global subscale | Baseline, end of treatment (at 3 weeks), 3-month follow-up
WOMAC physical function subscale | Baseline, end of treatment (at 3 weeks), 3-month follow-up
Overall pain measured on VAS | Baseline, end of treatment (at 3 weeks), 3-month follow-up
Hospital anxiety and depression scale | Baseline, end of treatment (at 3 weeks), 3-month follow-up
Aberdeen measure of participation | Baseline, end of treatment (at 3 weeks), 3-month follow-up
Mean analgesic intake per patient | Baseline, end of treatment (at 3 weeks), 3-month follow-up
Number of drop-outs because of adverse events | End of treatment (at 3 weeks), 3-month follow-up
Number of patients experiencing local adverse events | End of treatment (at 3 weeks), 3-month follow-up
Number of patients experiencing any side effects | End of treatment (at 3 weeks), 3-month follow-up
Number of patients experiencing serious side effects | End of treatment (at 3 weeks), 3-month follow-up
Number of drop-outs | End of treatment (at 3 weeks), 3-month follow-up
WOMAC pain subscale | Baseline, third treatment session, 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Reichenbach, MD, Principal Investigator — Institute of Social and Preventive Medicine (ISPM), University of Bern; Peter Jüni, Prof., Study Director — Applied Health Research Centre (AHRC), Li Ka Shing Knowledge Institute of St. Michael's Hospital, Department of Medicine and Institute of Health Policy, Management and Evaluation, University of Toronto, Canada
Locations (1):
- Institute of Social and Preventive Medicine (ISPM), University of Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Reichenbach S, Juni P, Hincapie CA, Schneider C, Meli DN, Schurch R, Streit S, Lucas C, Mebes C, Rutjes AWS, da Costa BR. Effect of transcutaneous electrical nerve stimulation (TENS) on knee pain and physical function in patients with symptomatic knee osteoarthritis: the ETRELKA randomized clinical trial. Osteoarthritis Cartilage. 2022 Mar;30(3):426-435. doi: 10.1016/j.joca.2021.10.015. Epub 2021 Nov 23. PMID 34826572